CLINICAL TRIAL: NCT04969120
Title: The Effect of Metoclopramide on the Length of First Stage of Labor in Nulliparous Women, a Randomized Controlled Trial
Brief Title: Metoclopramide and the Length of First Stage of Labor , a Randomized Controlled Trial
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Shaimaa Mostafa Mohammed Refaay El shemy, Lecturer of Obstetrics and gynecology at Cairo university, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: Metoclopramide and labour
Record Dates: First submitted 2021-06-27; First posted 2021-07-20 (Actual); Last update posted 2022-08-02 (Actual); Status verified 2022-08

CONDITIONS: Labour Duration and Metoclopramide
Keywords: Metoclopramide - labor duration-labor pain
MeSH Terms: interventions — Metoclopramide; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- (group 1) receiving intravenous metoclorpramide (Active Comparator): this group receive 10mg intravenous metoclopramide
  Interventions: Drug: Metoclopramide 10mg
- (group 2) receiving placebo (Placebo Comparator): this group receive 10mg intravenous placebo(0.9 sodium chloride)
  Interventions: Drug: Placebo (0.9 sodium chloride)

INTERVENTIONS:
Drug: Metoclopramide 10mg — this group receive 10mg intravenous metoclopramide slowly over 2 minutes the medication will be repeated every 2 hours for a maximum three doses
  Arms: (group 1) receiving intravenous metoclorpramide
Drug: Placebo (0.9 sodium chloride) — this group receive 10mg intravenous placebo(0.9 sodium chloride) slowly over 2 minutes the medication will be repeated every 2 hours for a maximum three doses
  Arms: (group 2) receiving placebo

SUMMARY:
Reducing the length of labor is a highly desirable goal of intrapartum care, both from a perspective of maternal and fetal well-being and for the providers of the birth services. Avoiding a long, protracted labor entails shorter exposure to pain anxiety and stress and would translate into a major improvement in maternal satisfaction with the childbirth experience.

Prolonged labor can lead to increased maternal and neonatal morbidity and mortality such as rupture of the uterus, postpartum hemorrhage, puerperal sepsis, and maternal death. Prolonged labor may be due to maternal age, premature rupture of membrane, epidural analgesia and the secretion of high levels of maternal stress hormones.

DETAILED DESCRIPTION:
Several studies showed that active management of labor could shorten the duration of labor, and the safety of this method has been demonstrated.

Metoclopramide binds to dopamine receptors acting as a receptor antagonist, and it is also a mixed serotonin receptor agonist and antagonist.

Metoclopramide could potentially reduce spasms of the smooth muscle of the cervix that remains richly innervated at birth and thus have a regulatory effect on cervical contractility, an interaction that might be important in aiding maximal tissue compliance, promoting cervical dilatation during labor, and helping to reduce dystocia. Dopamine and other catecholamines have been identified in rabbit, rat, guinea-pig, sheep, and human uteri.

The purpose of this study is to determine the effectiveness of metoclopramide for reducing the duration of spontaneous labor among nulliparous women managed according to a standard intrapartum protocol.

ELIGIBILITY:
Inclusion Criteria:

* primigravida
* singleton pregnancy
* termgestation (37-42 weeks)
* sure reliable dated
* vertex presentation , occipito-anterior position
* regular uterine contractions at every 5 minutes,each lasting for 20 seconds
* cervical dilatation of 5 cm
* with or without rupture of membrane
* no evidence of maternal or fetal distress

Exclusion Criteria:

* chorioamnionitis
* scarred uterus e.g. myomectomy
* cephalopelvic dispropotion
* history of cervical surgery or injury
* hypersensitivity to metoclopramide

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2022-07-01 (Actual)

PRIMARY OUTCOMES:
duration of labour | 8-12 hours
  cervical dilatation rate in first stage of labour

SECONDARY OUTCOMES:
labour pain | pain assessment at 30,60,120 minutes following injection of metoclopramide
  effect of metoclopramide on labour pain score using visual analogue scale which is a score from 0 to 10 cm The higher the score represents more pain

CONTACTS AND LOCATIONS:
Locations (1):
- Obstetrics and gynecology department at kasralainy hospital, Cairo, Egypt